CLINICAL TRIAL: NCT06547073
Title: Exploring the Possibilities of Virtual Reality in Rehabilitation of Patients With Frozen Shoulder
Brief Title: The Effect of Virtual Reality Training Compared to Traditional Exercise in Patients With Frozen Shoulder
Acronym: VR4shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2023-0381
Record Dates: First submitted 2024-06-18; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frozen shoulder group (Experimental): Patient group
  Interventions: Other: Virtual reality exercise training; Other: Traditional exercise training
- Healthy group (Active Comparator): Healthy subjects without shoulder pain
  Interventions: Other: Virtual reality exercise training

INTERVENTIONS:
Other: Virtual reality exercise training — Beat saber
Other: Traditional exercise training — Bench slides, supine active assisted flexion, pendulum exercise, seated active assisted external rotation
  Arms: Frozen shoulder group

SUMMARY:
Background: Virtual reality (VR) technology sees a rising appearance in clinical settings, and can be used for physical rehabilitation of the shoulder joint. The immersive virtual world created by VR games can be a distraction of the limitations and hindrances a patient experiences when exercising. Frozen shoulder (FS) or adhesive capsulitis is one of such instances of shoulder pathologies where pain and limited range of motion (ROM) are prev-alent and long lasting. VR could be an option to further help rehabilitate patients with FS.

Objectives: This study aims to investigate 3D upper limb kinematics of a FS patient during VR gaming and to compare these to the unaffected side, as well as to healthy participants. Additionally, this study also aims to compare the effects of a single session of VR gaming and traditional exercise training in patients with frozen shoulder on pain, ROM and shoulder strength as well as the participant's personal experience.

Study design: Cross sectional (3D kinematics) and randomized cross-over design (VR versus traditional exercise) Method: Patients with frozen shoulder (n=15) will be recruited through physical therapy practices and social media. Healthy subjects (n=30) will be recruited on social media. Both groups will play a VR game (Beat saber) will collecting 3D kinematic data of the upper limb with inertial measurement sensors (IMU's). Patients will be evaluated clinically before and after the VR session. The patient group will also perform a control intervention (traditional exercise program) and the same clinical evaluation will be performed before and after this session. Clinical evaluation will consist of shoulder range of motion measurment using a goniometer, pain evaluation using the visual analogue scale (VAS) and shoulder strength evaluation using a hand-held dynamometer (HHD). The order of sessions will be randomized for the patients. At the end of the study, both the healthy and patient group will be interviewed to report on their personal experiences with the VR intervention.

Outcome: 3D kinematics of the upper limb while playing a VR game will be compared between healthy and patient group to evaluate differences. In the patient group, the clinical effect of a single VR session will be compared to a single traditional exercise session.

ELIGIBILITY:
PATIENT GROUP (frozen shoulder

Inclusion Criteria:

* A diagnosis of frozen shoulder/adhesive capsulitis (by a medical doctor) both idiopathic and postoperative/posttraumatic
* The participants need to have:

  * a passive ROM restriction (measured using goniometry) at the affected shoulder of 25% or more in at least two directions in comparison to the unaffected shoulder
  * an external rotation restriction at the affected shoulder of at least 50% when compared to the unaffected side
  * pain and restricted ROM present for at least two months, reaching a plateau or becoming worse
  * gradual onset of pain and stiffness
* The participants are allowed to already be in therapy with a physiotherapist and do not have to stop an ongoing therapy in order to participate in the study. The reason for this is that only the short-term effect is being researched
* The participants are allowed to have had an operative treatment if they still have the aforementioned restrictions

Exclusion Criteria:

* The presence of contra-indications to perform active shoulder movements
* The presence of neurological conditions
* Systemic disease (e.g. Fibromyalgia, rheumatism, muscle disease…)
* The presence of visual conditions that will not allow performing VR therapy without losing balance
* A pathology of the back of lower limbs which do not allow the performance of exercise in standing position
* A higher risk of falling with at least one fall during the past year
* Insufficient control of the Dutch language

HEALTHY GROUP Exclusion criteria

* shoulder pain in the last 6 months
* prior shoulder surgery
* fractures of the upper arm or scapula
* systemic disease (e.g. Fibromyalgia, rheumatism, muscle disease…)
* the presence of contra-indications to perform active shoulder movements (e.g. recent elbow surgery), balance disorders (e.g. benign paroxysmal positional vertigo), visual disorders (e.g. severe reduced vision or visual acuity)
* any pathology in the back/lower limbs that prevents standing exercises from being performed
* increased risk of falls with at least one fall incident in the past year
* insufficient knowledge of the Dutch language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3D upper limb kinematics | During VR session (both groups) - Day 1
  Noraxon IMU

SECONDARY OUTCOMES:
Shoulder range of motion | Immediately before and after both interventions (patients group) - Day 1
  Goniometer
Shoulder strength | Immediately before and after both interventions (patients group) - Day 1
  Hand held dynamometer
Shoulder pain | Immediately before and after both interventions (patients group) - Day 1
  VAS
Personal experience with VR session | Immediately before and after both interventions (patients group) - Day 1
  Interview

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium